CLINICAL TRIAL: NCT06018610
Title: Mid-term Efficacy and Results of Postoperative Relaxation and Underfloor Classical Massage Methods and Training in Proximal Femur Fractures
Brief Title: Effectiveness of Relaxation and Massage Methods in Proximal Femur Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kalça kırığı
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Fracture of Femur
MeSH Terms: conditions — Femoral Fractures | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to conventional rehabilitation, relaxation exercises and classical massage of the sole of the foot will be applied to the study group. Patients will be re-evaluated 3 days after the completion of the interventions.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will receive conventional rehabilitation practices (in and out of bed strengthening exercises, for 3 days).
  Interventions: Other: Control

INTERVENTIONS:
Other: Rehabilitation — In addition to conventional rehabilitation, relaxation exercises and classical massage of the sole of the foot will be applied to the study group.
  Arms: Intervention Group
Other: Control — Conventional rehabilitation will be applied to the control group.
  Arms: Control Group

SUMMARY:
The study will be conducted with volunteer patients who are followed up by the Orthopedics and Traumatology Service of Muğla Sıtkı Koçman University Training and Research Hospital and who have undergone proximal femur fracture surgery and meet the study criteria. It is aimed to investigate the mid-term efficacy of relaxation exercises and classical massage of the sole of the foot applied in addition to the conventional physiotherapy program in the postoperative in-hospital period in patients with proximal femur fracture.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 50 years and older who were diagnosed with proximal femur fracture and underwent surgery
* No medical contraindications that would limit the ability to exercise
* Having a caregiver who can supervise the exercise program after discharge
* To be able to understand simple commands and to have signed the consent form

Exclusion Criteria:

* Patients with pathological fractures and/or multiple fractures
* Those with serious early complications
* Terminally ill patients
* Circumstances that would interfere with conducting assessments or communicating
* Lack of cooperation during the study
* Scoring ≤14 on the Mini Mental State Examinatio

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 3 days
  On a 10 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
Barthel Index (BI) | Change from Baseline BI at 3 days
  The Barthel Index was developed as a measure to assess disability in patients with neuromuscular and musculoskeletal disorders undergoing inpatient rehabilitation. A maximum total score of 100 can be obtained. Higher score indicates better condition.
EQ-5D-3L Quality of Life Scale | Change from Baseline EQ-5D-3L at 3 days
  The EQ-5D-3L provides information on three aspects of quality of life. Each dimension has three levels of impairment: no problems (level 1), some problems (level 2) and extreme problems (level 3). The score ranges from less than 0 to 1 (where 0 is a health status equivalent to death and negative values are worse than death) and 1 is the most positive score (the best perceived level according to the five dimensions included in the scale). Finally, the EQ VAS score is obtained by asking patients to rate their health status on a 20 cm vertical scale. The scale ranges from 0 to 100, with 0 meaning "worst imaginable health" and 100 meaning "best imaginable health".
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline HADS at 3 days
  The HADS consists of two subscales, one with seven items measuring anxiety and the other with seven items measuring depression, which are scored separately. Each item is answered by the patient on a 4-point response category (0 to 3), so that possible scores range from 0 to 21 for anxiety and 0 to 21 for depression. 0 to 7 is considered "normal", 8 to 10 "mild", 11 to 14 "moderate" and 15 to 21 "severe".
Tampa Scale for Kinesiophobia (TSK) | Change from Baseline TSK at 3 days
  The questionnaire is a 17-item scale developed to measure fear of movement/reinjury. The normal score range is between 17 and 68.
Nottingham Hip Fracture Score (NHFS) | Change from Baseline NHFS at 3 days
  The Nottingham Hip Fracture Score is an aggregate score of seven preoperative variables that gives an estimated risk of 30-day postoperative mortality using a standard logistic regression. This score is calculated based on age, gender, comorbidities, place of residence (i.e. home or institutional care), abbreviated mental test score (AMTS) and hemoglobin level at admission. Higher scores indicate better condition.
Sole sensory testing with Semmes-Weinstein Monofilament | Change from Baseline Semmes-Weinstein Monofilament Test at 3 days
  The filament is imposed horizontally against the skin until there is a visible bending of the fiber. The patient then verbally assesses whether the sensation is perceived. Starting with the thinnest filament, thick filament is used sequentially until the patient feels it.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet İmerci, MD, Study Director — Muğla Sıtkı Koçman University; Fatih Özden, PhD, Principal Investigator — Muğla Sıtkı Koçman University; Serkan Bakırhan, PhD, Principal Investigator — Ege University; İsmet Tümtürk, MSc, Principal Investigator — Süleyman Demirel University; Fatih Özyer, MD, Principal Investigator — Fethiye State Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Fethiye State Hospital, Muğla, Fethiye
  - Muğla Sıtkı Koçman Training and Research Hospital, Muğla, Menteşe

IPD SHARING:
Plan to Share IPD: No